CLINICAL TRIAL: NCT05262829
Title: A Single-arm, Open-label Clinical Study of Human Umbilical Cord Mesenchymal Stem Cells in the Treatment of Refractory Moderate to Severe Crohn's Disease
Brief Title: Clinical Study of Human Umbilical Cord Mesenchymal Stem Cells in the Treatment of Moderate and Severe Crohn's Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai East Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DFSC-2021(CR)-07
Record Dates: First submitted 2022-02-08; First posted 2022-03-02 (Actual); Last update posted 2023-02-17 (Actual); Status verified 2023-02

CONDITIONS: Crohn Disease
Keywords: Human Umbilical Cord Mesenchymal Stem Cells; Crohn Disease
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MSCs local treatment group/combined treatment group (Experimental): In the local treatment group, 60 million umbilical cord MSCs were injected into the diseased intestinal mucosa on the first day. In the combined treatment group, 60 million umbilical cord MSCs were injected into the diseased intestinal mucosa on the first day; on the second day, 1 million cells/kg of body weight were administered intravenously.
  Interventions: Biological: Human Umbilical Cord Mesenchymal Stem Cells

INTERVENTIONS:
Biological: Human Umbilical Cord Mesenchymal Stem Cells — MSCs treatment by intestinal submucosal injection/MSCs treatment by intravenous drip + MSCs treatment by intestinal submucosal injection

SUMMARY:
This is a prospective, single-arm, open-ended study to evaluate the efficacy and safety of human umbilical cord MSCs in the treatment of refractory moderate-to-severe Crohn's disease. The study protocol is either MSC injection into the patient's diseased intestinal mucosa or intravenous MSC injection + MSC injection into the patient's diseased intestinal mucosa. Follow-up time points were pre-treatment (week 0), week 4, week 8, week 12, and week 24 post-treatment, and the primary evaluation at follow-up was the number of subjects with clinical and endoscopic response or remission.

DETAILED DESCRIPTION:
This is a prospective, single-arm, open study to evaluate the efficacy and safety of human umbilical cord MSCs in the treatment of refractory moderate-to-severe Crohn's disease. The study will be conducted as follows: a total of 40 patients will be recruited and will receive either MSC injection into the diseased intestinal mucosa or intravenous MSC injection + MSC injection into the diseased intestinal mucosa. The proportion of patients with clinical and endoscopic response or remission will be used as the primary evaluation for follow-up. The Crohn's disease activity index (CDAI) was used to assess the severity of CD disease, with CDAI <150 considered to be in clinical remission; a decrease in CDAI ≥70 was considered to be clinically effective, also referred to as clinical response. Endoscopic response was defined as at least 50% improvement in the simplified endoscopic score for Crohn's disease (SES-CD) from baseline, and endoscopic remission was defined as a SES-CD score ≤2.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects aged between 18 and 70 years (including borderline values), of either sex.
2. Subjects with a comprehensive diagnosis of Crohn's disease for more than 3 months based on the patient's clinical presentation, endoscopy, imaging and pathology, with reference to the Consensus Opinion on the Diagnosis and Treatment of Inflammatory Bowel Disease in China (2018-Beijing).
3. Failure to respond to existing conventional therapy, or to primary or secondary treatment with TNF alpha monoclonal antibody, vedolizumab or ustekinumabd.
4. Current Crohn's disease with a Crohn's Disease Activity Index (CDAI) score ≥ 220 and ≤ 450.
5. Evidence of active inflammation and ulceration confirmed by endoscopy during screening.
6. Subjects must be free of active, latent, or undertreated Mycobacterium tuberculosis infection.
7. All women of childbearing potential and all men must be willing to use at least one highly effective method of contraception at the time of signing the consent form and throughout the study period until 1 month after the last dose of study drug.
8. Subjects who are willing and able to undergo treatment and follow-up, laboratory tests, and other study procedures as planned.
9. Subjects who are able to sign (and date) an informed consent form indicating that the subject has been informed of all relevant parts of the study
10. Subjects receiving non-disabling combination therapy for any reason must maintain a stable treatment regimen, defined as no stem cell therapy given or no dose change within 7 days or 5 half-lives (whichever is longer) prior to the initial stem cell injection.

Exclusion Criteria:

1. Presence of a complication of Crohn's disease, such as short bowel syndrome or any other manifestation that might be expected to require surgery, that prevents the use of CDAI to assess treatment response, or that might confound the assessment of the efficacy of MSC therapy.
2. Current abscess or suspected abscess. If the abscess has drained and been adequately treated 3 weeks prior to baseline (skin and perianal abscesses) and 8 weeks prior to baseline (intra-abdominal abscesses) then no exclusion is necessary. The prerequisite is that no further surgical treatment is anticipated. Subjects may be enrolled in the study if they have an active fistula that is not expected to require surgery and is confirmed to be abscess-free.
3. Subjects with evidence of pathogenic intestinal infection. Subjects with Clostridium difficile or other intestinal infections within 30 days of endoscopic screening, or subjects who screen positive for C. difficile toxin assay or other pathogens.
4. Subjects with total bilirubin, aspartate aminotransferase (AST) or alanine aminotransferase (ALT) above 2 times the upper limit of normal at the screening visit. Patients with cirrhosis will be excluded.
5. Subjects with eGFR ≤ 60 mL/min (as calculated by Cockcroft-Gault) or patients receiving hemodialysis.
6. Subjects with a current or clinically significant infection within 1 month prior to baseline, or history of more than one prior occurrence of herpes zoster, disseminated zoster (one occurrence) and other infections that the investigator believes may be exacerbated by participation in the study, or any infection requiring antimicrobial therapy within 2 weeks of screening.
7. Subjects who may currently be receiving any live virus vaccination or who have received any live virus vaccination within 8 weeks prior to baseline.
8. Subjects with a first-degree relative with a hereditary immunodeficiency.
9. History of any lymphoid proliferative disease (e.g., EBV-associated lymphoid proliferative disease), lymphoma, leukemia, myeloproliferative disease, multiple myeloma, or signs and symptoms suggestive of presenting lymphoid system disease.
10. Subjects who have received prior treatment with any lymphocyte depleting agent/therapy. Subjects with prior treatment with rituximab or other selective B lymphocyte depleting agents, but who have not received such treatment for at least 1 year prior to baseline, are eligible for the study.
11. Pregnant or lactating women or female subjects who are pregnant during planned enrollment in the study.
12. Prior history of alcohol or drug abuse and less than 6 months of abstinence prior to baseline.
13. Subjects with clinically relevant abnormalities confirmed by 12-lead ECG during the screening period that would affect their safety if enrolled in this study or affect the interpretation of the study results.
14. Subjects who have donated more than 500 mL of blood in the 2 months prior to baseline.
15. Subjects who have experienced major trauma or undergone major surgery within 4 weeks of the screening visit.
16. Subjects with a body temperature ≥38°C during the screening period or baseline period.
17. Subjects with malignancy or a history of malignancy.
18. Subjects infected with human immunodeficiency virus (HIV) or hepatitis B virus or hepatitis C virus.
19. Subjects who, in the opinion of the investigator, are uncooperative or unable to comply with the study procedures.
20. Any other condition that, in the opinion of the investigator, would render the subject unsuitable for enrollment in the study.
21. Subjects with preexisting or current clinically significant cardiovascular, neurological, psychiatric, renal, hepatic, immunological, gastrointestinal, genitourinary, neurological, musculoskeletal, cutaneous, sensory, endocrine (including uncontrolled diabetes or thyroid disease) or uncontrolled hematological abnormalities. "Clinically significant" is defined as a subject whose participation in the study would, in the opinion of the investigator, pose a risk to the safety of the subject or whose disease/condition would be exacerbated during the study in a manner that would affect the validity or safety analysis.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-02-28 (Actual); Primary Completion 2024-08-31 (Estimated); Study Completion 2025-01-31 (Estimated)

PRIMARY OUTCOMES:
Crohn's disease activity index score | Changes from baseline to week 4, week 8, week 12 and week 24 after stem cell treatment.
  The Crohn's Disease Activity Index (CDAI) was used to assess the severity of CD disease, and a CDAI <150 was considered clinically remitting; a decrease in CDAI ≥70 was considered clinically effective, also known as clinical response.
simplified endoscopic score for Crohn's disease | Changes from baseline to week 4, week 8, week 12 and week 24 after stem cell treatment.
  Endoscopic response was defined as at least 50% improvement in the simplified endoscopic score for Crohn's disease (SES-CD) from baseline, and endoscopic remission was defined as a SES-CD score ≤2.

SECONDARY OUTCOMES:
Inflammatory Bowel Disease Questionnaire | Changes from baseline to week 4, week 8, week 12 and week 24 after stem cell treatment.
  The Inflammatory Bowel Disease Questionnaire (IBDQ) is a widely used questionnaire for Health-related quality of life assessment in patients with inflammatory bowel diseases (IBDs).
Albumin | Changes from baseline to week 4, week 8, week 12 and week 24 after stem cell treatment.
  Albumin is an important component of the blood, and patients with severe Crohn's disease can present with clinical signs of hypoproteinemia.
Hemoglobin | Changes from baseline to week 4, week 8, week 12 and week 24 after stem cell treatment.
  Hemoglobin is an important component of the blood, and patients with severe Crohn's disease can present with clinical signs of anemia.
Fecal calprotectin | Changes from baseline to week 4, week 8, week 12 and week 24 after stem cell treatment.
  Fecal calprotectin (FC) is a non-invasive marker of gastrointestinal inflammation with advocated diagnostic precision in distinguishing inflammatory bowel disease (IBD) from non-IBD diagnoses.
body mass index (BMI) | Changes from baseline to week 4, week 8, week 12 and week 24 after stem cell treatment.
  Weight and height will be combined to report BMI in kg/m^2

CONTACTS AND LOCATIONS:
Overall Officials: Lan Zhong, MD, Study Director — Shanghai East Hospital
Locations (1):
- Shanghai East Hospital, Shanghai, Pudong New Area, China